CLINICAL TRIAL: NCT00341159
Title: Genetic Analysis of Cancer Susceptibility Alleles in the CARE Case-Control Study
Brief Title: Analysis of Data From the Women's Contraceptive and Reproductive Experiences (CARE) Study
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905089; 05-HG-N089
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-02-24

CONDITIONS: Breast Cancer
Keywords: Breast; BRCA1; BRCA2; Inherited; Association; Breast Cancer; Population-Based; Cancer Susceptibility Alleles
MeSH Terms: conditions — Breast Neoplasms

SUMMARY:
This study will continue to analyze data collected by the Women's Contraceptive and Reproductive Experiences (CARE) study. The CARE study was designed to evaluate the association between reproductive factors and risk of breast cancer in white and African-American women in the United States.

The present study is not recruiting additional participants. The original study enrolled 4,575 women with breast cancer and 4,682 control subjects between 35 and 64 years of age

All participants provided a blood sample for genetic study. The samples were analyzed for variants (mutations) in the BRCA1 and BRCA2 genes, the vitamin D receptor gene, the androgen receptor gene, and the insulin-like growth factor-1 gene.

In addition, all participants were interviewed to obtain information related to breast cancer risk, including a history of reproductive, menstrual, oral contraceptive, and hormone replacement therapy use; lifestyle factors such as smoking, alcohol use, body weight, and physical activity; history of medical conditions and procedures; demographic characteristics, such as age, race, marital status, and so forth; and a detailed family history of cancer.

DETAILED DESCRIPTION:
The purpose of the women's CARE study was a population based case control study designed to evaluate risk factors for breast cancer among white and African American women ages 35-64 in the United States. The study cases were U.S. born English-speaking women newly diagnosed with pathologically confirmed invasive breast cancer between July 1994 and April 1998. Cases were identified by the Surveillance, Epidemiology and End Results (SEER) cancer registry at each center except for Philadelphia where they were ascertained by field staff from local hospitals. African-American women were over sampled, as were younger case patients to maximize numbers in those strata. Older white case patients were randomly sampled to provide approximately equal numbers of patients in each 5-year age category. A total of 4575 cases were interviewed including 2953 white women and 1622 African American women.

Controls were U.S. born English-speaking women who had never been diagnosed with invasive or in situ breast cancer identified by random digit dialing. Controls were frequency-matched to cases by study center, race, and five-year age group. A total of 4682 controls were interviewed of which 3021 were white and 1661 were African American.

Information collected similarly from cases and controls focused on factors potentially related to the risk of breast cancer, including, reproductive, menstrual, oral contraceptive (OC) and Hormone Replacement Therapy (HRT) use histories; lifestyle factors such as smoking, alcohol use, body weight, and physical activity; selected history of medical conditions and procedures; demographic characteristics; and a detailed family history of cancer.

A total of 1652 Cases and 1453 controls provided high quality DNA in the form of blood samples. The Ostrander lab's role in the study was to screen the complete coding region, as well as intron-exon boundaries of 1652 cases and 600 controls for mutations in the BRCA1 and BRCA2 genes using both denaturing high performance liquid chromatograph (DHPLC) and direct sequencing. In addition we screened 1652 cases and 1453 controls for germline variants in the androgen receptor (AR), Insulin Like Growth Factor-1 (IGF-1) and vitamin D receptor (VDR) genes. The lab work for the study has been completed, and analysis is currently underway. This IRB file does not include a request to do any additional lab work. The focus of this request is to continue analysis of the now completed lab work in collaboration with the data-coordinating center at the Fred Hutchinson Cancer Research Center. Data coordination is lead by Drs. Kathleen Malone and Janet Daling of the Public Health Sciences Division of the FHCRC.

ELIGIBILITY:
* Original recruitment were cases identified by the Surveillance, Epidemiology and End Results (SEER) cancer registry several years ago for the data set. Accrual is now completed.

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9257 (Actual)
Dates: Start 2005-01-18; Study Completion 2015-02-24

CONTACTS AND LOCATIONS:
Overall Officials: Elaine A Ostrander, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hall JM, Lee MK, Newman B, Morrow JE, Anderson LA, Huey B, King MC. Linkage of early-onset familial breast cancer to chromosome 17q21. Science. 1990 Dec 21;250(4988):1684-9. doi: 10.1126/science.2270482.
- [Background] Narod SA, Feunteun J, Lynch HT, Watson P, Conway T, Lynch J, Lenoir GM. Familial breast-ovarian cancer locus on chromosome 17q12-q23. Lancet. 1991 Jul 13;338(8759):82-3. doi: 10.1016/0140-6736(91)90076-2. PMID 1676470
- [Background] Wooster R, Neuhausen SL, Mangion J, Quirk Y, Ford D, Collins N, Nguyen K, Seal S, Tran T, Averill D, et al. Localization of a breast cancer susceptibility gene, BRCA2, to chromosome 13q12-13. Science. 1994 Sep 30;265(5181):2088-90. doi: 10.1126/science.8091231.